CLINICAL TRIAL: NCT05947032
Title: Effects of Supervised Endurance Training Versus Home-based Exercise Plan on Functional Capacity and Fatigue Among Pulmonary Arterial Hypertension Patients
Brief Title: Supervised Endurance Training Among Pulmonary Arterial Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01603 Farheen Khan
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised endurance exercise training + Patient Education (Experimental)
  Interventions: Other: Supervised endurance exercise training + Patient Education
- Home exercises + Patient Education (Active Comparator)
  Interventions: Other: Home exercises + Patient Education

INTERVENTIONS:
Other: Supervised endurance exercise training + Patient Education — ENDURANCE TRAINING:
  Treadmill Walking:
  Frequency: 15 to 20 sessions for 3 to 5 days per week. Intensity: 40% to 60% of HRR Time: 15 Min Type: aerobic training
  Recumbent Bike:
  Frequency: 15 to 20 sessions for 3 to 5 days/week. Intensity: 40% to 60% HRR Time: 15 Min Type: aerobic training
  + Patient Education
  Arms: Supervised endurance exercise training + Patient Education
Other: Home exercises + Patient Education — HOME EXERCISES:
  CONVENTIONAL Treatment:
  Walking:
  Frequency: 2 times/ day Intensity: as tolerated Time: 30 Min Type: aerobic training
  Stair climbing:
  Frequency: 1 flight/ day Type: aerobic training
  + Patient Education
  Arms: Home exercises + Patient Education

SUMMARY:
To compare the effects of supervised endurance training versus home based exercise plan on functional capacity and fatigue among pulmonary arterial hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary arterial hypertension, not pregnant and tobacco free.
* Age = 21 to 82
* Patients with documented PAH diagnosed by echocardiography (enlarged RA an enlarged RV with a thick wall, septal shift by enlarged chambers of right side of heart, an elevated mPAP) or a resting mean pulmonary arterial pressure equal to 25mm Hg determined by right heart catheterization.
* Patients on stable PH therapies, sedentary, and had no pulmonary rehabilitation for 6 months prior to enrolment.

Exclusion Criteria:

* Patients will be excluded if they are not able to complete 6MWT.
* A documented pulmonary capillary wedge pressure greater then or equal to 15 mm Hg.
* Significant hepatic, renal, metabolic or mitochondrial dysfunctions; severe psychiatric disease; use of beta-adrenergic blockers or antiretroviral therapies; and any musculoskeletal or neurological condition that would limit walking or exercise performance.
* Patients with a history of heart failure.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 4 weeks
  It measures the patient's perception of the influence of fatigue on physical and social functioning through patient's response to nine different question. Scoring is based on likert scale where 1 indicates strong agreement and 7 indicates strong disagreement. A score of 4 or greater is indicative of severe fatigue.
Human Activity Profile | 4 weeks
  A questionnaire to assess the activity level of patient in rehabilitation with a total no of 94 questions I ascending order based on metabolic demands. For each activity mentioned patient will be asked 1) if they are still doing this activity 2) have stopped doing this activity or never did this activity. HAP generates two scores the maximum activity score MAS and adjusted activity score ASS. Score < 53 is considered as low activity score between 54-73 stands for intermediate activity for high activity score > 74 is required respectively.
6MWT Distance | 4 weeks
  Subject walks as fast as they can for 6 mins on a walking track to determine their ability to participate in physical activity.The 6 MWT is scored as the total distance covered in the 6-min duration of the test. it will be measured in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No